CLINICAL TRIAL: NCT00062712
Title: Induction of Donor Specific Immunologic Hyporesponsiveness With Thymoglobulin, Sirolimus and Donor Bone Marrow Infusion
Brief Title: Evaluating the Use of Thymoglobulin, Sirolimus, and Donor Bone Marrow With Kidney Transplantation Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030204; 03-DK-0204
Record Dates: First submitted 2003-06-11; First posted 2003-06-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-22

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression; Transplant; Kidney Transplant
MeSH Terms: interventions — Antilymphocyte Serum; Sirolimus

INTERVENTIONS:
Drug: Allogeneic Bone Marrow, Anti-Thymocyte Globulin (Sangstat) & Sirolimus (Wyeth-Ay

SUMMARY:
Patients with renal failure need chronic dialysis or a kidney transplant to survive. Most kidney transplant patients must take medicines indefinitely to prevent their immune systems from rejecting the kidney. Long-term exposure to these anti-rejection medicines can damage the transplanted kidney.

The purpose of this study is to determine whether giving patients cells from the donor's bone marrow will reduce or eliminate the need for long-term use of these anti-rejection drugs. In addition to the donor's bone marrow cells, patients will receive the drugs thymoglobulin and sirolimus.

A total of 20 patients will participate in this five-year study.

DETAILED DESCRIPTION:
This protocol will evaluate the combination of Thymoglobulin (Sangstat), sirolimus and donor bone marrow infusion for its ability to induce a state of donor specific hematopoietic chimerism and immune hyporesponsiveness within the context of renal transplantation. Thymoglobulin (Sangstat), a FDA-approved polyclonal rabbit-IgG antithymocyte preparation, will be given for up to ten days at the time of transplantation to effect lymphocyte depletion. This will be combined with sirolimus (rapamycin, Wyeth-Ayerst), an oral immunosuppressant agent recently approved by the FDA. Sirolimus allows for antigen specific T cell activation but prevents T cell clonal expansion by interrupting IL-2 receptor beta-chain signal transduction. Donor bone marrow will be administered seven days following transplant. Patients demonstrating six months of rejection free graft survival will have their sirolimus withdrawn over three months beginning at the sixth month anniversary of the transplant.

Twenty people will be evaluated in this pilot protocol. Approximately ten will receive living donor kidney allografts and the remaining patients will receive cadaveric kidney allografts. Patients will be treated with Thymoglobulin beginning prior to graft implantation and continuing for approximately ten days. Glucocorticosteroids will be given during the first Thymoglobulin treatment to limit monocyte activation and prevent the cytokine release syndrome associated with the initial administration of this antibody preparation. Patients will be given sirolimus orally beginning the day after transplantation and continuously thereafter. Donor bone marrow will be administered seven days following transplantation. Patients will then be monitored for evidence of allograft rejection using standard functional parameters and protocol allograft biopsies. In addition, patients will be followed for specific desired effects, including a transient state of donor hematopoietic mixed microchimerism and allospecific AICD. Both of these are expected to promote the development of allospecific graft tolerance. This will be accomplished by assaying peripheral blood and allograft biopsies for apoptosis and the peripheral blood for evidence of alloreactive T cell clone depletion and donor chimerism.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates for a kidney transplant.

Age 12 through 60 at the time of transplant for the first 10 patients transplanted. Age 12 through 75 for subsequent patients. Patients younger than age 12 are better served being transplanted in a center with more extensive pediatric medical and nephrology support. Patients less than 12 years of age are also at higher risk for post transplant lymphoproliferative disorder following transplant than adults and intensive induction immunosuppression increases the risk further. The use of aggressive induction imunosuppression in this population would be inappropriate. Patients over the age of 75 generally require less immunosuppression than younger patients. The use of aggressive induction immunosuppression in this population would be inappropriate.

Willingness to give informed consent.

Availability of donor tissue for testing. This could include splenic or peripheral blood lymphocytes from a cadaveric donor or a willing living donor enrolled on the Clinical Center Living Donor Protocol who consents to periodic phlebotomy for peripheral blood lymphocyte isolation.

Availability of adequate donor bone marrow for infusion.

EXCLUSION CRITERIA:

Immunosuppressive drug therapy at the time of or 2 months prior to enrollment. Specifically, candidates may not be taking prednisone, cyclosporine, tacrolimus, azathioprine, mycophenolate mofetil, antilymphocyte agents, cyclophosphamide, methotrexate, or other agents whose therapeutic effect is immunosuppressive.

Treatment with a nucleoside analogue chemotherapeutic agent (i.e. fludarabine phosphate, cladribine, or pentostatin) within 12 months of kidney transplant.

Absolute lymphocyte count less than 1000/mm(3) prior to first dose of Thymogobulin.

Any active malignancy or any history of a hematologic malignancy or lymphoma. Patients with primary, cutaneous basal cell or squamous cell cancers may be enrolled providing the lesions are appropriately treated prior to transplant.

Donor/recipient combinations in which there are 0 HLA mismatches or in which the donor is homozygous for a shared HLA haplotype. Serologic HLA typing to be conducted at the Walter Reed Army Medical Center Tissue Typing Laboratory.

Sensitization as defined by historical or current PRA less than 20 percent in patients receiving their first kidney allograft.

First kidney graft survival less than 3 years as a consequence of acute/chronic rejection or positive T or B cell crossmatch in patients receiving second kidney allograft.

Historical or current positive T cell cross match between donor and recipient.

Significant coagulopathy or requirement for anticoagulation therapy that would contraindicate protocol allograft biopsies.

Platelet count less than 75,000/mm(3) at the time of transplant.

Any known immunodeficiency syndrome such as HIV, Chronic Granulomatous Disease, Severe Combined Immunodeficiency, DiGeorge Syndrome, etc.

Presence of uncorrected cardiac insufficiency (either valvular or vascular) or major vascular disease.

Subjects unwilling/unable to practice birth control if potentially fertile.

Presence of active or chronic infection.

Any condition that would likely increase the risk of protocol participation or confound data interpretation such as inability or unwillingness to comply with protocol monitoring and therapy, including, among others, a history of noncompliance, circumstances where compliance with protocol requirements is not feasible due to living conditions, travel restrictions, access to urgent medical services, or access to anti-rejection drugs after the research protocol is completed.

Any history of allergy or anaphalaxis to rabbit proteins.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2003-06-09; Study Completion 2007-03-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wilson M, Burt AR, Milligan G, Anderson NG. Wortmannin-sensitive activation of p70s6k by endogenous and heterologously expressed Gi-coupled receptors. J Biol Chem. 1996 Apr 12;271(15):8537-40. doi: 10.1074/jbc.271.15.8537. PMID 8621477